CLINICAL TRIAL: NCT02979093
Title: Oxytocin and Brain Reward and Stress Responses to Infant Cues in Addicted Mothers
Brief Title: Oxytocin and Brain Responses in Maternal Addiction
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to recruit proposed study sample size due to COVID restrictions.
Sponsor: Lane Strathearn, MBBS PhD (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor-Investigator, Lane Strathearn, MBBS PhD, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 201601749
Record Dates: First submitted 2016-11-17; First posted 2016-12-01 (Estimated); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Maternal Behavior; Maternal Addiction
Keywords: maternal drug addiction; mother-infant attachment; intranasal oxytocin; unresolved trauma; maternal brain responses; mother-infant synchrony
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Addicted (Other): The addiction group will be scanned twice using functional magnetic resonance imaging (fMRI). Subjects will be randomly assigned to receive either the active comparator (intranasal oxytocin spray) or the placebo comparator before the first scanning session. For the second scan (approximately one month later), the subject will receive the other spray which she did not receive at the time of the first scan.
  Interventions: Drug: Oxytocin; Drug: Placebos; Procedure: Functional MRI scanning
- Control (Other): The control group will be scanned twice using functional magnetic resonance imaging (fMRI). Subjects will be randomly assigned to receive either the active comparator (intranasal oxytocin spray) or the placebo comparator before the first scanning session. For the second scan (approximately one month later), the subject will receive the other spray which she did not receive at the time of the first scan.
  Interventions: Drug: Oxytocin; Drug: Placebos; Procedure: Functional MRI scanning

INTERVENTIONS:
Drug: Oxytocin — All women will receive a nasal spray containing oxytocin.
  Other Names: Pitocin; Syntocinon
Drug: Placebos — All women will receive a nasal spray containing a placebo solution.
Procedure: Functional MRI scanning — Study participants undergo two functional MRI scans.

SUMMARY:
A prior study by the principal investigator of this project identified dopamine- and oxytocin-related brain pathways that showed a diminished response when addicted mothers viewed the faces of their own vs. unknown infants, compared with non-addicted mothers. These areas include the hypothalamus, striatum and ventromedial prefrontal cortex. In addition, the investigators plan to examine activation patterns within the salience network, which includes the anterior cingulate cortex and the anterior insula. Oxytocin, a neuropeptide with decreased blood levels seen in addicted mothers, is integrally involved in maternal brain and behavioral responses. When administered intranasally, the pilot data has shown enhanced activation of the striatum, prefrontal cortex (PFC) and amygdala.

The purpose of this study is to continue and expand upon the previous investigation of maternal addiction, by conducting a randomized, double-blinded, placebo controlled, crossover study of intranasal oxytocin on maternal brain responses. 150 mothers from the University of Iowa and the Yale Child Study Center will be enrolled (75 with a history of drug addiction and 75 matched control mothers), along with their 2 to 12-month-old infants, to participate in four study visits over a two-month period.

DETAILED DESCRIPTION:
Maternal drug addiction constitutes a major public health problem for both women and affected children, with long lasting consequences on children's social, emotional and cognitive development. Current treatment strategies tend to focus on the mother and her current addiction, rather than her relationship with her child, and developmental processes that may perpetuate the addiction problems, such as unresolved childhood attachment trauma, neglect, and chronic stress. Unlike mothers who find engaging with their own infant to be a uniquely rewarding experience, mothers with addictions may be less able to respond appropriately to their infant's cues, finding them less intrinsically rewarding or salient, and more stress provoking.

Aim 1: To examine, in addicted mothers compared to non-addicted control mothers, the effect of intranasal oxytocin (OT) on functional MRI brain responses to reward-related cues: own vs. unknown happy infant faces.

Aim 2: To examine, in addicted mothers compared to non-addicted control mothers, the effect of intranasal OT on brain responses to stress-related cues: own vs. unknown sad infant faces and cries.

Aim 3: To examine the effect of intranasal OT on functional brain connectivity, including the striatum, PFC and amygdala. Specifically, exploring whether, after receiving intranasal OT compared to placebo, addicted mothers show increased functional connectivity between the amygdala and (i) the ventromedial PFC for own-happy infant faces, and (ii) the dorsolateral PFC and striatum for own-sad faces.

Aim 4: To explore how individual differences in adult attachment and mother-infant synchrony, sensation-seeking/risk-taking and stress/trauma exposure are associated with OT brain responses to infant faces.

Aim 5: To examine the effect of intranasal OT on activation of the salience network in addicted mothers, as well as connectivity patterns between these regions and the amygdala. We predict that there will be noticeable increase in activity in the salience network (dorsal anterior cingulate and anterior insula) after administering OT. We predict the addiction group will have a greater affect from the OT treatment than the control group.

ELIGIBILITY:
Inclusion Criteria for addiction sample:

Drug-addicted subjects will be English speaking adult women who:

1. are being evaluated for treatment of their addiction or are currently enrolled in treatment programs;
2. have an infant <12 months;
3. meet criteria for substance abuse or dependence in the past year, as assessed by MINI International Neuropsychiatric Interview (MINI);
4. have a substance abuse history, including use during the most recent pregnancy;
5. are recommended at intake for drug-treatment services for substance abuse;
6. are 18 years to 40 years old; and
7. have been speaking English or enrolled in English-speaking school since age 8.

Inclusion Criteria for non-addicted mothers (controls):

Control subjects will be English-speaking adult women who:

1. have an infant <12 months of age;
2. do not meet criteria for past or present drug abuse or dependence;
3. are 18 years to 40 years old; and
4. have been speaking English or enrolled in English-speaking school since age 8.

Exclusion Criteria for addiction sample:

Potential drug-addicted subjects will be ineligible if they have:

1. severe psychiatric or substance-related symptoms requiring in-patient psychiatric hospitalization or detoxification for suicidality, homicidality, grave disability, physiological alcohol or drug withdrawal within the last 30 days;
2. past or present diagnosis of schizophrenia or other psychotic disorders;
3. metal implants or other contraindications for MRI scanning;
4. pending legal cases (e.g., outstanding arrest warrants or parental rights hearings) prohibiting them from completing the study;
5. current pregnancy or plans to become pregnant during the course of the study;
6. infants with clinical evidence of in utero drug effects, such as opiate withdrawal symptoms during the neonatal period, facial dysmorphism or intrauterine growth restriction (IUGR) or microcephaly;
7. infants with birth weight less than 3 lb. 5 oz.;
8. infants who have significant vision, hearing or motor problems (such as cerebral palsy) that cannot be corrected;
9. mothers who have significant vision or hearing problems that cannot be corrected;
10. out-of-home placement of infant for the past month or more than 50% of child's life;
11. delivered more than one baby during most recent pregnancy (twins, triplets, etc.).
12. exclusively breastfeeding

Exclusion criteria for non-addicted mothers:

Potential control subjects will be ineligible if they have:

1. positive drug toxicology screen at any point in the study;
2. drug abuse or dependence based on MINI in the past year or lifetime;
3. use of tobacco products in the past 2 years;
4. current hazardous alcohol use as ascertained by AUDIT score > 8;
5. present or past history of ambulatory detoxification;
6. severe psychiatric symptoms requiring inpatient psychiatric hospitalization for suicidality, homicidality, grave disability, physiological alcohol or drug withdrawal within the past 30 days;
7. past or present diagnosis of schizophrenia or other psychotic disorders;
8. metal implants or other contraindications for MRI scanning;
9. current pregnancy or plans to become pregnant during the course of the study;
10. infants with birth weight less than 3 lb. 5 oz.;
11. infants who have significant vision, hearing or motor problems that cannot be corrected (such as cerebral palsy);
12. mothers who have significant vision or hearing problems that cannot be corrected;
13. out-of-home placement of infant for the past month or more than 50% of child's life; and
14. delivered more than one baby during most recent pregnancy (twins, triplets, etc.).
15. exclusively breastfeeding

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lane Strathearn, MBBS PhD, Principal Investigator — University of Iowa; Linda Mayes, MD, Principal Investigator — Yale University; Helena Rutherford, PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale Child Study Center, New Haven, Connecticut
  - University of Iowa, Iowa City, Iowa

IPD SHARING:
Plan to Share IPD: No
The University of Iowa and Yale will compile data from both sites for data analysis purposes only. There is no plan to make individual participant data available.

REFERENCES:
- [Background] SAMHSA, "Results from the 2011 National Survey on Drug Use and Health: Summary of National Findings" (Substance Abuse and Mental Health Services Administration, Rockville, MD, 2012).
- [Background] Chaffin M, Kelleher K, Hollenberg J. Onset of physical abuse and neglect: psychiatric, substance abuse, and social risk factors from prospective community data. Child Abuse Negl. 1996 Mar;20(3):191-203. doi: 10.1016/s0145-2134(95)00144-1. PMID 8734549
- [Background] Rutherford HJ, Williams SK, Moy S, Mayes LC, Johns JM. Disruption of maternal parenting circuitry by addictive process: rewiring of reward and stress systems. Front Psychiatry. 2011 Jul 6;2:37. doi: 10.3389/fpsyt.2011.00037. eCollection 2011. PMID 21779252
- [Background] Strathearn L, Li J, Fonagy P, Montague PR. What's in a smile? Maternal brain responses to infant facial cues. Pediatrics. 2008 Jul;122(1):40-51. doi: 10.1542/peds.2007-1566. PMID 18595985
- [Background] Kim S, Fonagy P, Allen J, Strathearn L. Mothers' unresolved trauma blunts amygdala response to infant distress. Soc Neurosci. 2014;9(4):352-63. doi: 10.1080/17470919.2014.896287. Epub 2014 Mar 17. PMID 24635646
- [Background] L. C. Mayes, R. Feldman, R. Granger, The effects of polydrug use with and without cocaine on mother infant interaction at 3 and 6 months. Infant behavior & development 20, 489 (1997).
- [Background] Strathearn L, Mayes LC. Cocaine addiction in mothers: potential effects on maternal care and infant development. Ann N Y Acad Sci. 2010 Feb;1187:172-83. doi: 10.1111/j.1749-6632.2009.05142.x. PMID 20201853
- [Background] Strathearn L, Mertens CE, Mayes L, Rutherford H, Rajhans P, Xu G, Potenza MN, Kim S. Pathways Relating the Neurobiology of Attachment to Drug Addiction. Front Psychiatry. 2019 Nov 8;10:737. doi: 10.3389/fpsyt.2019.00737. eCollection 2019. PMID 31780957

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 59 participant mothers were enrolled in this component of the study. Their infants did not participate in the scanning sessions or receive oxytocin/placebo sprays and were not considered enrolled in this portion of the study. 11 mothers did not participate in scanning session, leaving 48 mothers who participated in the first scanning session. 43 mothers had 74 usable scanning sessions (31 with 2 sessions [62 sessions], and 12 with one session).
Units Other Than Participants: Scans
Groups:
- ADDICTION: PLACEBO FIRST GROUP: The addiction group participants are scanned twice using functional magnetic resonance imaging (fMRI). These participants receive the placebo comparator before the first scanning session, and the active comparator (intranasal oxytocin spray) before the second scanning session (approximately one month later).
- ADDICTION: OXYTOCIN FIRST GROUP: The addiction group will be scanned twice using fMRI. These participants receive active comparator (intranasal oxytocin spray) before the first scanning session, and the placebo comparator before the second scanning session (approximately one month later).
- CONTROL: PLACEBO FIRST GROUP: The control group participants are scanned twice using fMRI. These participants receive the placebo comparator before the first scanning session, and the active comparator (intranasal oxytocin spray) before the second scanning session (approximately one month later).
- CONTROL: OXYTOCIN FIRST GROUP: The control group will be scanned twice using fMRI. These participants receive active comparator (intranasal oxytocin spray) before the first scanning session, and the placebo comparator before the second scanning session (approximately one month later).
Period: First Scan Session
Arm/Group | ADDICTION: PLACEBO FIRST GROUP | ADDICTION: OXYTOCIN FIRST GROUP | CONTROL: PLACEBO FIRST GROUP | CONTROL: OXYTOCIN FIRST GROUP
Started | 12; 12 Scans | 12; 12 Scans | 12; 12 Scans | 12; 12 Scans
Completed (Scanning session with usable data.) | 11; 11 Scans | 10; 10 Scans | 10; 10 Scans | 12; 12 Scans
Not Completed | 1; 1 Scans | 2; 2 Scans | 2; 2 Scans | 0; 0 Scans
Not completed — Scanning data problems | 1 | 2 | 2 | 0
Period: Second Scan Session
Arm/Group | ADDICTION: PLACEBO FIRST GROUP | ADDICTION: OXYTOCIN FIRST GROUP | CONTROL: PLACEBO FIRST GROUP | CONTROL: OXYTOCIN FIRST GROUP
Started (The number of participants in the "Second Scan Session" is not equal to the number who completed the "First Scan Session" because some participants without usable data from the first session still completed the Second Scan Session.) | 9; 9 Scans | 7; 7 Scans | 11; 11 Scans | 11; 11 Scans
Completed (Scanning session with usable data) | 6; 6 Scans | 7; 7 Scans | 10; 10 Scans | 8; 8 Scans
Not Completed | 3; 3 Scans | 0; 0 Scans | 1; 1 Scans | 3; 3 Scans
Not completed — Scanning data problems | 3 | 0 | 1 | 3

BASELINE CHARACTERISTICS:
Population: 11 of these participants did not complete any scanning visits (5 addiction, 6 controls), and thus were not assigned to an Arm.
Groups:
- Addicted Mothers: The addiction group will be scanned twice using functional magnetic resonance imaging (fMRI). Subjects will be randomly assigned to receive either the active comparator (intranasal oxytocin spray) or the placebo comparator before the first scanning session. For the second scan (approximately one month later), the subject will receive the other spray which she did not receive at the time of the first scan.
  Oxytocin: All mothers will receive a nasal spray containing oxytocin.
  Placebos: All mothers will receive a nasal spray containing a placebo solution.
  Functional MRI scanning: Study mothers undergo two functional MRI scans.
  Infants did not participate in scanning sessions, so baseline measures are not reported.
- Control Mothers: The control group will be scanned twice using functional magnetic resonance imaging (fMRI). Subjects will be randomly assigned to receive either the active comparator (intranasal oxytocin spray) or the placebo comparator before the first scanning session. For the second scan (approximately one month later), the subject will receive the other spray which she did not receive at the time of the first scan.
  Oxytocin: All mothers will receive a nasal spray containing oxytocin.
  Placebos: All mothers will receive a nasal spray containing a placebo solution.
  Functional MRI scanning: Study mothers undergo two functional MRI scans.
  Infants did not participate in scanning sessions, so baseline measures are not reported.
- Total: Total of all reporting groups
Arm/Group | Addicted Mothers | Control Mothers | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Categorical [Count of Participants; unit: Participants] — Maternal age at Visit 1.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 29 | 30 | 59
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Maternal age at Visit 1.
  years | 29.3 (6.8) | 29.0 (4.8) | 29.1 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Only includes mothers, and not their infants.
  Participants
    Female | 29 | 30 | 59
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 27 | 29 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 25 | 29 | 54
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Effect of Intranasal Oxytocin on Brain fMRI Activation, Independent of Addiction Status (Hypotheses 1 and 2A).
Description: Brain activation (blood-oxygen level dependent [BOLD] signal) in response to reward-related cues (own [O] vs. unknown [U] infant happy faces).
  Brain activation (BOLD signal) in response to stress-related cues (own [O] vs. unknown [U] infant sad faces).
  Specific regions of interests include the striatum and amygdala (for both happy and sad faces).
Time Frame: 50 minutes after administration of oxytocin or placebo
Population: Sample consists of both mothers with addiction and mothers who have no history of addiction, with one or two scanning sessions. Individuals with movement artifact or preprocessing problems removed. As pre-specified in the study protocol and similar to most functional MRI studies, the contrasts between two stimuli are reported (e.g., own vs unknown baby faces).
Measure: Least Squares Mean (Standard Error); unit: BOLD signal
Units Other Than Participants: Number of Scanning sessions
Groups:
- Oxytocin; Placebo: Each participant will be scanned twice using functional magnetic resonance imaging (fMRI). Subjects will be randomly assigned to receive either the active comparator (intranasal oxytocin spray) or the placebo comparator before the first scanning session. For the second scan (approximately one month later), the subject will receive the other spray which she did not receive at the time of the first scan.
  Oxytocin: All women will receive a nasal spray containing oxytocin.
  Placebos: All women will receive a nasal spray containing a placebo solution.
  Functional MRI scanning: Study participants undergo two functional MRI scans.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 34 | 40
Number analyzed (Number of Scanning sessions) | 34 | 40
BOLD signal
  Happy faces (O>U): Striatum | -.33 (.16) | .00678 (.14)
  Happy faces (O>U): Amygdala | -.25 (.16) | .16 (.15)
  Sad faces (O>U): Striatum | .34 (.14) | .04 (.13)
  Sad faces (O>U): Amygdala | .36 (.14) | .04 (.13)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; This analysis is for Striatum: Happy Own vs. Happy Unknown; Test type: Superiority; p = 0.106, Mixed Models Analysis — Unadjusted; Mean Difference (Final Values) = 0.1697, Standard Error of Mean 0.1025
Statistical Analysis 2: Comparison: Oxytocin vs Placebo; This analysis is for the Amygdala: Happy Own vs. Happy Unknown infant faces; Test type: Superiority; p = 0.0709, Mixed Models Analysis — Unadjusted; Mean Difference (Final Values) = 0.20458, Standard Error of Mean 0.11010
Statistical Analysis 3: Comparison: Oxytocin vs Placebo; This analysis is for Striatum: Sad Own vs. Sad Unknown infant faces; Test type: Superiority; p = 0.0964, Mixed Models Analysis — Unadjusted; Mean Difference (Final Values) = -0.14559, Standard Error of Mean 0.08546
Statistical Analysis 4: Comparison: Oxytocin vs Placebo; This analysis is for Amygdala: Sad Own vs. Sad Unknown infant faces; Test type: Superiority; p = 0.0538, Mixed Models Analysis — Unadjusted; Mean Difference (Final Values) = -0.15755, Standard Error of Mean 0.07914

2. Primary Outcome: Effect of Intranasal Oxytocin on Brain fMRI Activation in Addicted vs Controls Mothers (Hypotheses 1 and 2B)
Description: Brain activation (BOLD signal) in response to reward-related cues (own [O] vs. unknown [U] infant happy faces). Specific region of interest includes the ventromedial prefrontal cortex (vmPFC) (interaction effect).
  Brain activation (BOLD signal) in response to stress-related cues (own vs. unknown infant sad faces). Specific region of interest includes the dorsolateral prefrontal cortex (dlPFC) (interaction effect).
Time Frame: 50 minutes after administration of oxytocin or placebo
Population: The fMRI data was obtained from 43 participant mothers (21 in the Addiction group and 22 in the Control group), each of whom provided one or two valid scanning session, totaling 74 sessions. Of the 21 Addiction mothers, 15 contributed scanning data in the Oxytocin condition, and 19 in the Placebo condition. Of the 22 Control mothers, 19 contributed data in the Oxytocin condition, and 21 in the Placebo condition. As pre-specified in the protocol, the contrasts between two stimuli are reported.
Measure: Least Squares Mean (Standard Error); unit: BOLD signal
Units Other Than Participants: Scanning session
Groups:
- Addicted - Oxytocin Condition: The addiction group will be scanned twice using functional magnetic resonance imaging (fMRI). Subjects will be randomly assigned to receive either the active comparator (intranasal oxytocin spray) or the placebo comparator before the first scanning session. For the second scan (approximately one month later), the subject will receive the other spray which she did not receive at the time of the first scan.
  Oxytocin: All women will receive a nasal spray containing oxytocin.
  Functional MRI scanning: Study participants undergo two functional MRI scans.
- Control - Oxytocin Condition: The control group will be scanned twice using functional magnetic resonance imaging (fMRI). Subjects will be randomly assigned to receive either the active comparator (intranasal oxytocin spray) or the placebo comparator before the first scanning session. For the second scan (approximately one month later), the subject will receive the other spray which she did not receive at the time of the first scan.
  Oxytocin: All women will receive a nasal spray containing oxytocin.
  Functional MRI scanning: Study participants undergo two functional MRI scans.
- Addicted - Placebo Condition: The addiction group will be scanned twice using functional magnetic resonance imaging (fMRI). Subjects will be randomly assigned to receive either the active comparator (intranasal oxytocin spray) or the placebo comparator before the first scanning session. For the second scan (approximately one month later), the subject will receive the other spray which she did not receive at the time of the first scan.
  Placebo: All women will receive a nasal spray containing placebo.
  Functional MRI scanning: Study participants undergo two functional MRI scans.
- Control - Placebo Condition: The control group will be scanned twice using functional magnetic resonance imaging (fMRI). Subjects will be randomly assigned to receive either the active comparator (intranasal oxytocin spray) or the placebo comparator before the first scanning session. For the second scan (approximately one month later), the subject will receive the other spray which she did not receive at the time of the first scan.
  Placebos: All women will receive a nasal spray containing a placebo solution.
  Functional MRI scanning: Study participants undergo two functional MRI scans.
Arm/Group | Addicted - Oxytocin Condition | Control - Oxytocin Condition | Addicted - Placebo Condition | Control - Placebo Condition
Number analyzed (Participants) | 15 | 19 | 19 | 21
Number analyzed (Scanning session) | 15 | 19 | 19 | 21
BOLD signal
  Happy faces (O>U): vmPFC | .00266 (0.20) | -0.30 (0.18) | 0.20 (0.18) | -0.11 (0.18)
  Sad faces (O>U): dlPFC | 0.48 (0.20) | 0.39 (0.19) | 0.06 (0.19) | -0.02 (0.18)
Statistical Analysis 1: Comparison: Addicted - Oxytocin Condition vs Control - Oxytocin Condition vs Addicted - Placebo Condition vs Control - Placebo Condition; This is a mixed effects model with group (Addiction vs. Control) and condition (Oxytocin [OT] vs Placebo). Both variables were included in the model. The interaction effect was tested but not included in the model. This result focuses on OT vs. placebo for Ventromedial prefrontal cortex (vmPFC) for happy own vs. happy unknown infant faces; Test type: Superiority; p = 0.319, Mixed Models Analysis — unadjusted; Mean Difference (Final Values) = 0.09778, Standard Error of Mean 0.09687
Statistical Analysis 2: Comparison: Addicted - Oxytocin Condition vs Control - Oxytocin Condition vs Addicted - Placebo Condition vs Control - Placebo Condition; This is a mixed effects model with group (addiction vs. control) and condition (OT vs Placebo). Both variables were included in the model. The interaction effect was tested but not included in the model. This result focuses on addiction vs. control for vmPFC for Happy Own vs. Happy Unknown infant faces; Test type: Superiority; p = 0.171, Mixed Models Analysis — unadjusted; Mean Difference (Final Values) = -0.15289, Standard Error of Mean 0.10968
Statistical Analysis 3: Comparison: Addicted - Oxytocin Condition vs Control - Oxytocin Condition vs Addicted - Placebo Condition vs Control - Placebo Condition; This is a mixed effects model with group (addiction vs. control) and condition (OT vs Placebo). Both variables were included in the model. The interaction effect was tested but not included in the model. This result focuses on OT vs placebo for Dorsolateral Prefrontal Cortex (dlPFC) for Sad Own vs. Sad Unknown infant faces; Test type: Superiority; p = 0.0179, Mixed Models Analysis — Unadjusted; Mean Difference (Final Values) = -0.20839, Standard Error of Mean 0.08405
Statistical Analysis 4: Comparison: Addicted - Oxytocin Condition vs Control - Oxytocin Condition vs Addicted - Placebo Condition vs Control - Placebo Condition; This is a mixed effects model with group (addiction vs. control) and condition (OT vs Placebo). Both variables were included in the model. The interaction effect was tested but not included in the model. This result focuses on addiction vs. control for dlPFC for Sad Own vs. Sad Unknown infant faces; Test type: Superiority; p = 0.7171, Mixed Models Analysis — unadjusted; Mean Difference (Final Values) = 0.04315, Standard Error of Mean 0.11827

ADVERSE EVENTS:
Time Frame: Approximately 4-6 months.
Description: Infants did not participate in scanning sessions, so adverse events were not collected.
Groups:
- ADDICTION: PLACEBO: This arm includes the addiction group during the scanning session under the placebo condition.
- ADDICTION: OXYTOCIN: This arm includes the addiction group during the scanning session under the oxytocin condition.
- CONTROL: PLACEBO: This arm includes the control group during the scanning session under the placebo condition.
- CONTROL: OXYTOCIN: This arm includes the control group during the scanning session under the oxytocin condition.
Arm/Group | ADDICTION: PLACEBO | ADDICTION: OXYTOCIN | CONTROL: PLACEBO | CONTROL: OXYTOCIN
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT02979093/Prot_SAP_000.pdf